CLINICAL TRIAL: NCT00444522
Title: Safety, Tolerability, and Pharmacokinetics of a Single Dose of StaccatoTM Alprazolam for Inhalation in Normal, Healthy Volunteers
Brief Title: Staccato Alprazolam Single Dose PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexza Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMDC-002-101
Record Dates: First submitted 2007-03-05; First posted 2007-03-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2007-03

CONDITIONS: Healthy
Keywords: Panic attacks, Staccato® Alprazolam
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Alprazolam thermal aerosol

SUMMARY:
We are developing Staccato Alprazolam for the acute treatment of panic attacks associated with panic disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 to 55 years, inclusive.
2. Subjects with a body mass index (BMI) ≥21 and ≤30.
3. Subjects who speak, read, and understand English and are willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures.
4. Subjects who are willing and able to be confined to the Clinical Research Unit (CRU) and comply with the study schedule and study requirements.
5. Subjects who are in good general health as determined by a complete medical history, physical examination, 12-lead ECG, spirometry, blood chemistry profile, hematology, and urinalysis.

Exclusion Criteria:

1. Subjects who regularly consume large amounts of xanthine-containing substances (ie, more than 5 cups of coffee or equivalent amounts of xanthine-containing substances per day).
2. Subjects who have taken prescription or nonprescription medication (with the exception of vitamins and acetaminophen if medically necessary) within 5 days of Visit 2 (Baseline).
3. Subjects who have had an acute illness within 5 days of Visit 2 (Baseline).
4. Subjects who have received an investigational drug within 30 days (or within 5 half lives investigational drug, if >30 days) prior to Visit 2 (Baseline).
5. Subjects who have smoked tobacco within the last year.
6. Subjects who have a history within the past 2 years of drug or alcohol dependence or abuse as defined by DSM-4.
7. Subjects with a history of HIV positivity.
8. Subjects with a history of allergy or intolerance to benzodiazepines or related drugs (alprazolam, lorazepam, diazepam, etizolam, clonazepam, adinazolam).
9. Subjects who test positive for alcohol or have a positive urine drug screen at Visit 1 or Visit 2.
10. Subjects who have hypotension (systolic blood pressure ≤90 mmHg, diastolic blood pressure ≤50 mmHg), or hypertension (systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥90 mmHg).
11. Subjects who have a clinically significant ECG abnormality.
12. Subjects with a history of unstable angina, syncope, coronary artery disease, myocardial infarction, congestive heart failure (CHF), stroke, transient ischemic attack (TIA), or a neurological disorder.
13. Subjects who have a history of pulmonary disease that precludes administration of Staccato Alprazolam (asthma, bronchitis, bronchospasm, emphysema).
14. Subjects who have an FEV1 less than 80% of predicted values on spirometry assessments at Visit 1.
15. Female subjects who are breastfeeding or have a positive pregnancy test at Visit 1 or Visit 2.
16. Female participants of child-bearing potential or within 1 year of menopause, and sexually active are excluded unless they use a medically acceptable and effective birth control method throughout the study and for 1 week following the end of the study. Medically acceptable methods of contraception include abstinence, diaphragm with spermicide, intrauterine device (IUD), condom with foam or spermicide, vaginal spermicidal suppository, surgical sterilization, and progestin implant or injection. Unacceptable methods include: birth control pills, patches, and injections, the rhythm method, withdrawal, condoms alone, or diaphragm alone.
17. Subjects who have any other disease or condition, by history, physical examination, or laboratory abnormalities that in the investigator's opinion, would present undue risk to the subject, or may confound the interpretation of study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2005-06 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile and dose proportionality

CONTACTS AND LOCATIONS:
Overall Officials: Randall Stoltz, MD, Principal Investigator — West Pharmaceutical Services, GFI Research Center, Evansville, IN 47714

IPD SHARING:
Plan to Share IPD: Yes
IPD submitted to regulatory authorities. Others may contact Alexza Pharmaceuticals, Inc. Please send your request to ClinicalTrialsInfo@alexza.com